CLINICAL TRIAL: NCT04606238
Title: Preference-based Decision Aid to Support Participatory Decisions About Tumor-specific and Palliative Therapy in the Last Months of Life
Brief Title: Decision Aid to Support Advanced Cancer Patients
Acronym: PETUPAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other); Heidelberg University (Other); University of Jena (Other); Bielefeld University (Other)
Responsible Party: Principal Investigator, Eva Winkler, Prof. Dr. med. Dr. phil. Director of the NCT-EPOC Programme (Ethics and Patient oriented Care) at the National Center for Tumor Diseases, University Hospital Heidelberg
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: UHHeidelberg
Record Dates: First submitted 2020-10-06; First posted 2020-10-28 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Advanced Cancer
Keywords: decision aid; advanced cancer; forgoing of cancer treatment; patients' inclusion in clinical trials; pre-post design study
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group without DA (No Intervention): adult patients with incurable, stage IV disease (Prostate-, Breast-, Pancreatic-, Stomach- and Colorectal cancer) in an advanced treatment stage.
- Group with DA (Other): adult patients with incurable, stage IV disease (Prostate-, Breast-, Pancreatic-, Stomach- and Colorectal cancer) in an advanced treatment stage.
  Interventions: Other: Decision Aid

INTERVENTIONS:
Other: Decision Aid — Oncologists and patients will use the decision aid in the same situation (change of treatment needs to be discussed with the patient - either because of disease progression or treatment toxicity or other reasons (e.g. change of care setting).
  Arms: Group with DA

SUMMARY:
To support advanced cancer patients, for whom standard therapy is no longer available, and their oncologists in therapy decisions, the investigators aim to develop a decision-making aid (DA) in a multi-phased bicentric study. The DA aims to help patients to understand better risks and benefits of available treatment options including the options of standard palliative care, off-label drug use within an individual treatment plan and involvement in early clinical trials.

DETAILED DESCRIPTION:
Decisions about the provision of anticancer therapy and the initiation of palliative care in the last months of life are frequent and challenging in clinical practice. Research indicates that there is considerable heterogeneity regarding clinical practice in this context and that oncologists' values influence treatment decisions, as well as whether or not patients participate in these decisions. While there is evidence that seriously ill patients differ in their choices between treatment options compared to healthy persons, as well as in their evaluation of treatment goals and related care settings, there is a lack of analysis regarding criteria relevant to patients in the last 6 months of life, when assessing the benefit of anticancer treatment and palliative care. Yet, in decisions about anticancer treatment and involvement of palliative care, patients' preferences and values are of particular importance since anticancer treatment - while associated with high expectations for a positive effect - often has only marginal influence on prognosis towards the end of a cancer trajectory and sometimes forestalls choosing a palliative care setting or coping with the disease. Hence, the decision has a high impact on patients' last months of life. Involving patients more actively in the planning of their care has been on the agenda for more than a decade, but the implementation of this idea in routine clinical practice remains a challenge. Instead, oncologists often avoid prognosticating and eliciting patient preferences for or against anticancer treatment and values in the last phase of life. One important reason is that oncologists report discussions about ending anticancer therapy the most challenging communication task.

To support advanced cancer patients, for whom standard therapy is no longer available, and their oncologists in therapy decisions, the investigators aim to develop a decision-making aid (DA) in a multi-phased bicentric study. The DA aims to help patients to understand better risks and benefits of available treatment options including the options of standard palliative care, off-label drug use within an individual treatment plan and involvement in early clinical trials.

Methods and analysis:

In phase I, the DA will be developed after exploration of decisional needs of patients and views of health care providers based on face-to face interviews and focus groups discussions. Subsequently, the DA will be alpha-tested and redrafted, as necessary, in phase II. In phase III, the DA will be (1) beta-tested with patients and oncologists and (2), and assessed by experts. In the last project phase, the investigators will run a pre-post design study with doctor-patient-encounters to access improvements on primary study outcome, i.e. patients' level of decisional conflict. In addition, the user acceptance will be tested.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* adult patients with incurable, stage IV disease in an advanced treatment stage (prognosis <12 months and/or standard palliative care);
* adequate level of German language;
* willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Patients that already are under standard palliative care only;
* are cognitive impaired;
* have extreme anxiety or distress;
* have a severe comorbid illness excluding antitumor treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Level of decisional conflict | Baseline
  Level of decisional conflict will be measured with the Decision Conflict Scale that assesses patients' perceptions of uncertainty, modifiable factors con-tributing to uncertainty, and ultimate satisfaction with the choice. It is one of the most robust and validated instruments to test the impact of decision aids also in end-of-life decision making. It has 16 items and 5 response categories, ranging from "0" -strongly agree till "4"-strongly disagree
Level of decisional conflict | 26 weeks
  Level of decisional conflict will be measured with the Decision Conflict Scale that assesses patients' perceptions of uncertainty, modifiable factors con-tributing to uncertainty, and ultimate satisfaction with the choice. It is one of the most robust and validated instruments to test the impact of decision aids also in end-of-life decision making. It has 16 items and 5 response categories, ranging from "0" -strongly agree till "4"-strongly disagree

SECONDARY OUTCOMES:
Patients' involvement in decision-making | Baseline
  Patients' involvement in decision-making will be assessed with the German questionnaire on shared decision making. It has 9 items with 6-points Likert scale, ranging from "0-not at all" till "6 -fully correct". The higher score means more shared decision making.
Patients' involvement in decision-making | 26 weeks
  Patients' involvement in decision-making will be assessed with the German questionnaire on shared decision making. It has 9 items with 6-points Likert scale, ranging from "0-not at all" till "6 -fully correct". The higher score means more shared decision making.
The trade-off between patients' preferences for quality and length of life | Baseline
  The trade-off between patients' preferences for quality and length of life will be assessed with the German validated version of "Quality and Quantity Questionnaire" The questionnaire consists of nine items in two preference dimensions: Q(uality) of life (QL) and L(ength) of life (LL).
  Patients indicate how strongly they agree or disagree with the statements on a 5-point Likert scale. High scores on the quantity or quality scale indicate the importance of length or quality of life, respectively.
The trade-off between patients' preferences for quality and length of life | 26 weeks
  The trade-off between patients' preferences for quality and length of life will be assessed with the German validated version of "Quality and Quantity Questionnaire" The questionnaire consists of nine items in two preference dimensions: Q(uality) of life (QL) and L(ength) of life (LL).
  Patients indicate how strongly they agree or disagree with the statements on a 5-point Likert scale. High scores on the quantity or quality scale indicate the importance of length or quality of life, respectively.
Preferred role of the patient in decision-making | Baseline
  Preferred role of the patient in decision-making will be assessed with a German version of the Control Preference Scale (CPS). It consists of five statement (A, B, C, D, E) that each portrays a different role in treatment decision-making. For analysis a categorical variable, which is the person's most preferred role in treatment decision-making, will be created. Preference orders will be reclassified into Active (A, B), Collaborative ( C) and Passive (D, E). Ordinal categorical analysis can be applied.
Preferred role of the patient in decision-making | 26 weeks
  Preferred role of the patient in decision-making will be assessed with a German version of the Control Preference Scale (CPS). It consists of five statement (A, B, C, D, E) that each portrays a different role in treatment decision-making. For analysis a categorical variable, which is the person's most preferred role in treatment decision-making, will be created. Preference orders will be reclassified into Active (A, B), Collaborative ( C) and Passive (D, E).Ordinal categorical analysis can be applied.
Satisfaction with the oncologist-patient interaction | Baseline
  Satisfaction with the oncologist-patient interaction will be assessed using the validated questionnaire on the Quality of Physician-Patient Interaction (QQPPI). It has 14 Items with a 5-point scale (range: 1 [I do not agree] to 5 [I fully agree]).
Satisfaction with the oncologist-patient interaction | 26 weeks
  Satisfaction with the oncologist-patient interaction will be assessed using the validated questionnaire on the Quality of Physician-Patient Interaction (QQPPI). It has 14 Items with a 5-point scale (range: 1 [I do not agree] to 5 [I fully agree]).
Effect on hope | Baseline
  Effect on hope will be assessed with a German Version of the Herth Hope Index (HHI-D). It has 12 items with a 4-point Likert scale. Higher scores indicate more hope.
Effect on hope | 26 weeks
  Effect on hope will be assessed with a German Version of the Herth Hope Index (HHI-D). It has 12 items with a 4-point Likert scale. Higher scores indicate more hope.
Effect on patients' quality of life | Baseline
  Quality of life will be assessed with the EORTC QLQ-C30, a questionnaire developed to measure the quality of life of cancer patients. The QLQ-C30 has global health status, five functional scales, and three symptom scales. High scores of functional scales means healthy functioning. A high score for global health status means a higher quality of life. A high score of symptom scales demonstrates a high level of problems. Scores for all scales and single items range from 0 to 100.
Effect on patients' quality of life | 26 weeks
  Quality of life will be assessed with the EORTC QLQ-C30, a questionnaire developed to measure the quality of life of cancer patients. The QLQ-C30 has global health status, five functional scales, and three symptom scales. High scores of functional scales means healthy functioning. A high score for global health status means a higher quality of life. A high score of symptom scales demonstrates a high level of problems. Scores for all scales and single items range from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Laryionava K, Schildmann J, Wensing M, Wedding U, Surmann B, Woydack L, Krug K, Winkler E. Development and Evaluation of a Decision Aid to Support Patients' Participatory Decision-Making for Tumor-Specific and Palliative Therapy for Advanced Cancer: Protocol for a Pre-Post Study. JMIR Res Protoc. 2021 Sep 17;10(9):e24954. doi: 10.2196/24954. PMID 34533464